CLINICAL TRIAL: NCT02406222
Title: Pomalidomide in Relapsed and Refractory Multiple Myeloma (RRMM)
Acronym: MUKseven
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM13/10758
Record Dates: First submitted 2015-02-18; First posted 2015-04-02 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory; Pomalidomide; Dexamethasone; Cyclophosphamide
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomalidomide and Dexamethasone (Active Comparator): Pomalidomide and Dexamethasone will be administered as part of a 28 day cycle. Patients will continue with their treatment until disease progression, intolerance, toxicity or withdrawal.
  Dosing schedule:
  * Pomalidomide 4mg orally on days 1-21
  * Dexamethasone 40mg orally on days 1, 8, 15 and 22
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide Dexamethasone Cyclophosphamide (Experimental): Pomalidomide, Dexamethasone and Cyclophosphamide will be administered as part of a 28 day cycle. Patients will continue with their treatment until disease progression, intolerance, toxicity or withdrawal.
  Dosing schedule:
  * Pomalidomide 4mg orally on days 1-21
  * Dexamethasone 40mg orally on days 1, 8, 15 and 22
  * Cyclophosphamide 500mg orally on days 1, 8 and 15
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pomalidomide — Chemotherapy
Drug: Dexamethasone — Chemotherapy
Drug: Cyclophosphamide — Chemotherapy
  Arms: Pomalidomide Dexamethasone Cyclophosphamide

SUMMARY:
This study is determining whether the addition of cyclophosphamide to pomalidomide and dexamethasone improves progression free survival in patients with relapsed refractory myeloma (RRMM) compare to pomalidomide and dexamethasone alone. Patients will be randomised on a 1:1 basis to receive CPD or Pd. Treatment will be continued until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Multiple myeloma is the second most common hematologic malignancy in the European Union (EU), responsible for an estimated 21,000 deaths in the EU in 2008. For patients that relapse or are refractory to current standard treatment (combination of bortezomib/lenalidomide, dexamethasone and an alkylating agent) there are few options available and therefore the prognosis within this group is often poor with response to treatment decreasing with successive relapses until resistant disease develops. . Current standard treatment at first relapse in the UK is the use of bortezomib in combination with dexamethasone and cyclophosphamide. Another common treatment is lenalidomide given with dexamethasone and cyclophosphamide. The addition of cyclophosphamide has demonstrated to improve treatment outcomes whilst being tolerated well. A recent clinical study has shown the addition of cyclophosphamide to the combination of pomalidomide and dexamethasone has shown to be safe and tolerable and beneficial in terms of treatment outcomes. The primary aim of this study is to investigate whether the addition of cyclophosphamide to pomalidomide and dexamethasone leads to an improved progression free survival. A secondary aim is to identify markers from clinical material that will predict response to pomalidomide in a group of relapsed and refractory multiple myeloma (RRMM) patients to provide important information for use in discussions with NICE on how best to improve the value and use of pomalidomide in the UK in the RRMM setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic multiple myeloma (according to International Myeloma Working Group (IMWG) 2009 criteria) and have measurable disease
* Participants must require therapy for relapsed and/or refractory disease
* Participants must have received ≥ 2 treatment lines of anti-myeloma therapy (induction therapy followed by autologous stem-cell transplantation (ASCT) and consolidation/maintenance will be considered as one line).
* Participants must have received prior treatment with both lenalidomide and proteasome inhibitor, either as single agents or in combination regimens
* All participants must have failed treatment with either lenalidomide and proteasome inhibitor in one of the following ways:

  1. Documented progressive disease on or within 60 days of completing treatment with lenalidomide and/or proteasome inhibitor ; or
  2. In case of prior response [≥ partial response (PR)] to lenalidomide or proteasome inhibitor, participants must have relapsed within 6 months after stopping treatment with lenalidomide and/or proteasome inhibitor containing regimens; or
  3. Participants who have not had a ≥ minimal response (MR) despite receiving at least 4 cycles of treatment or who have developed intolerance/toxicity after a minimum of two cycles of lenalidomide and/or proteasome inhibitor containing regimen
* Patients must have received adequate prior alkylator therapy in one of the following ways

  1. As part of a stem cell transplant; or
  2. A minimum of 4 consecutive cycles of an alkylator based therapy; or
  3. Progression on treatment with an alkylator; provided that the participant received at least 2 cycles of an alkylator containing therapy.
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Required laboratory values within 14 days of treatment:

  * Absolute neutrophil count ≥ 1.0 x109 /L (growth factor support is permitted)
  * Platelet count ≥ 30 x 109/L (platelet transfusion is permitted)
  * Creatinine clearance > 30 mL/min
  * Corrected serum calcium ≤ 3.5 mmol/L
  * Haemoglobin ≥ 8 g/dL (blood transfusion support is permitted)
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) < 3 times Upper Limit of Normal (ULN)
  * Serum total bilirubin < 17 µmol/l
* Participants must consent to provide the bone marrow samples specified at screening and throughout the trial, in order to enter the trial. Confirmation of receipt of the sample from the lab must be received before treatment commences..
* Able to give informed consent and willing to follow trial protocol
* Aged over 18 or over
* Females of childbearing potential (FCBP) must agree to utilise one reliable form of contraception for 28 days prior to starting trial treatment, during the trial, and for 28 days after trial treatment discontinuation and even in the case of dose interruption and must agree to regular pregnancy testing during this timeframe
* Females must agree to abstain from breastfeeding during trial participation and 28 days after trial drug discontinuation
* Males must agree to use a latex condom during any sexual contact with FCBP during the trial, including during any dose interruptions and for 28 days following discontinuation from this trial even if he has undergone a successful vasectomy
* Males must also agree to refrain from donating semen or sperm while on pomalidomide, including during any dose interruptions and for 28 days after discontinuation from this trial
* All participants must agree to refrain from donation blood while on trial drug, including during dose interruptions and for 28 days after discontinuation from this trial

Exclusion Criteria:

* Previous therapy with pomalidomide
* Hypersensitivity to thalidomide, lenalidomide, cyclophosphamide or dexamethasone
* Participants with non-secretory multiple myeloma
* Peripheral neuropathy ≥ Grade 3
* Participants who have received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant
* Participants who are planned for a stem cell transplant post MUK Seven trial treatment
* Antitumour therapies including investigational medicinal products at any dose within 28 days before the start of protocol treatment (or 5 half-lives, whichever is longer). Bisphosphonates for bone disease and radiotherapy for palliative intent are permitted.
* Participants with any of the following

  1. Uncontrolled congestive heart failure
  2. Myocardial infarction within 12 months prior to starting trial treatment
  3. Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
* Participants with gastrointestinal disease that may significantly alter absorption of pomalidomide
* Participants with a history of other malignancies within 5 years before the date of study entry (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that is considered cured with minimal risk of recurrence within 5 years).
* Participants unable or unwilling to undergo antithrombotic prophylactic treatment
* Pregnant or breastfeeding females
* Participants known to be seropositive for HIV, or active infectious hepatitis A, B or C
* Any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From randomisation up to 72 months
  To determine whether the addition of cyclophosphamide to pomalidomide and dexamethasone (CPD) improves progression-free survival in patients with relapsed refractory myeloma (RRMM) in the UK, compared to pomalidomide and dexamethasone (Pd) alone

SECONDARY OUTCOMES:
Maximum response overall | From the start of treatment up to 72 months
  To determine the maximum response achieved from treatment
Response to treatment | From the start of treatment up to 72 months
  Determine the response to treatment
Clinical benefit rate overall | From the start of treatment up to 72 months
  Determine any clinical benefit that is derived from treatment
Time to maximum response | From the start of treatment up to 72 months
  Determine the time to maximum response to treatment
Duration of response | From the start of treatment up to 72 months
  Determine the duration that the response to treatment lasts for
Overall survival | Date of randomisation to death, up to 72 months
  Determine overall survival for all patients that receive treatment
Treatment compliance | From the start of treatment up to end of treatment
  Measured by treatment delays and missed treatment doses
Safety and Toxicity | Time of registration to 28 days post treatment discontinuation
  Measured by adverse reactions and serious adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaiser, Dr, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (21):
- United Kingdom (21):
  - Belfast Health & Social Care Trust, Belfast
  - University of Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Queens Hospital, Burton-on-Trent
  - University Hospital of Wales NHS Trust, Cardiff
  - Ninewells Hospital, Dundee
  - Beatson Oncology Centre, Glasgow
  - St James's Hopsital, Leeds
  - University Hospital of Leicester NHS Trust, Leicester
  - St Bartholomew Hospital, London
  - University College London Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College Hospital, London
  - Central Manchester Univeristy Hospital NHS Trust, Manchester
  - The Christie Hospital, Manchester
  - Churchill Hospital, Oxford
  - Sheffield Teaching Hospitals NHS FoundationTrust, Sheffield
  - University Hospital of North Tees, Stockton-on-Tees
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No